CLINICAL TRIAL: NCT05413408
Title: Chinese Culture-Specific Intervention to Decrease the Stigma of Nursing Students Towards Schizophrenia--A Pilot Randomized Controlled Trial
Brief Title: Intervention to Decrease the Stigma of Nursing Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HSEARS20220127002
Record Dates: First submitted 2022-05-25; First posted 2022-06-10 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2022-03

CONDITIONS: Stigma, Social
MeSH Terms: conditions — Social Stigma | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- education and contact to change participants stigma towards schizophrenia (Experimental): The intervention consists of three phases, including investigative learning activity (this section will last about one week), higher-order thinking activity (this section will last about two hours), collaborative activity (this section will last about two hours). Both the intervention group and the control group will be interns in the hospital simultaneously. The study outcomes include nursing students' knowledge, attitude, and behavioral intentions regarding stigma towards schizophrenia. The intervention effect will be evaluated by the researcher, comparing results between and within the two groups from baseline (T0) to immediately after first and second session intervention (T1), immediately after third session intervention (T2), and three months follow-up (T3).
  Interventions: Other: Education and contact
- Participants reading a book about schizophrenia knowledge (Active Comparator): The control group only has one session and will be given a book of schizophrenia knowledge, and they will be asked to finish reading it in four weeks.
  Interventions: Other: Education and contact

INTERVENTIONS:
Other: Education and contact — The intervention consists of three phases, including investigative learning activity (this section will last about one week), higher-order thinking activity (this section will last about two hours), collaborative activity (this section will last about two hours). Both the intervention group and the control group will be interns in the hospital simultaneously. The study outcomes include nursing students' knowledge, attitude, and behavioral intentions regarding stigma towards schizophrenia. The intervention effect will be evaluated by the researcher, comparing results between and within the two groups from baseline (T0) to immediately after first and second session intervention (T1), immediately after third session intervention (T2), and three months follow-up (T3).
  The control group only has one session and will be given a book of schizophrenia knowledge, and they will be asked to finish reading it in four weeks.

SUMMARY:
not

DETAILED DESCRIPTION:
Introduction Mental illness stigma is influenced by empathy, culture, and beliefs. However, few researchers specifically consider empathy, culture, and beliefs when designing interventions to reduce stigma. Schizophrenia is the most stigmatized mental illnesses. Nursing students will play the role of health educators and provide care for patients in the future. Their stigmas will negatively impact the care quality provided to people diagnosed with schizophrenia if not properly attended. This study intends to examine the feasibility, acceptability, and preliminary efficacy of an education and contact intervention programme aiming to improve nursing students' knowledge and empathy of schizophrenia and decrease their negative attitudes and stigma behavior towards people with schizophrenia. Methods and Analysis This is a two-phase study design. Phase 1 development includes a literature review and a descriptive qualitative study. Phase 2 is a pilot study, the feasibility, accessibility, and efficacy of the pilot RCT will be assessed by the quantitative and qualitative study. In the first phase, descriptive qualitative study with focus group and a literature review will be used to inform the intervention development of a pilot RCT. The second phase includes a pilot RCT including 60 nursing students who 7 practice in clinical settings of a tertiary hospital. These nursing students will be randomly assigned into the intervention group and the control group. The pilot study intervention consists of three stages, including the investigative learning activity (lasting about 6 hours), the collaborative activity (lasting about 4 hours), and the higher-order thinking activity (lasting about 4 hours). Both the intervention group and the control group will be interns in the tertiary hospital simultaneously when they take part in this study. The control group go through only one stage--they will be given a book about schizophrenia knowledge and asked to finish reading it in four weeks. After the pilot intervention study, there will be a process evaluation of a qualitative interview. Both first and second phase qualitative study will use qualitative research of fourth-year nursing students being focus groups interviewed. The pilot intervention study outcomes include nursing students' knowledge, attitude, and behavioral intentions regarding stigma towards schizophrenia, and nursing students' empathy towards people with schizophrenia. The pilot intervention study effect will be evaluated by the researcher and the results of the two groups will be compared on the baseline (T0), post-intervention (T1), and three months follow-up (T2).

ELIGIBILITY:
Inclusion Criteria:

* Participants should be 18 years old or above.
* Participants should complete all the school courses to ensure that they have similar theoretical knowledge in psychiatric nursing.
* Participants can communicate in Mandarin.
* Participants are voluntarily participating in this study.
* Participants have not participated in any other similar intervention before.
* Participants are doing a clinical practicum in Xiangya Hospital, Changsha, Hunan Province.

Exclusion Criteria:

* Participants are receiving treatment of schizophrenia or other mental illness.
* Participants are lack of essential equipment to take an online interview.
* Regular personal contact with someone with schizophrenia or other mental illness (more than three times a month). Because people's prejudice may decrease when they meet and interact with people with mental illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Subject recruitment time | up to one month
  The time used for subject recruitment
Achievable recruitment rate | up to one month
  the ratio between the number of nursing students actually participating and the number of potential nursing students that need to participat
Eligibility rate of participants | up to one month
  the number of participants eligible for this study/number of participants screened prior to eligibility assessment.
The response rate of scales | up to three month
  the proportions of missing values on the items of each scale
Drop-out rate of participants | up to three month
  the number of nursing students who drop out in each intervention session to the number of intervention groups

SECONDARY OUTCOMES:
Knowledge of Schizophrenia as assessed by Knowledge about Schizophrenia Test (KAST) | up to three month
  Knowledge about Schizophrenia Test (KAST)-Chinese version will be used to measure the stigma-related schizophrenia knowledge of participants. KAST, including 18 items, demonstrate an acceptable reliability coefficient of 0.68. The content validity index of items (I-CVI) ranged from 0.83 to 1.00, while the S-CVI/UA and S-CVI/Ave were 0.83 and 0.97, respectively, and known-group validity was satisfactory.
Attitudes of Schizophrenia as assessed by Mental Illness Clinicians' Attitudes Scale (MICA) | up to three month
  Mental Illness Clinicians' Attitudes Scale (MICA)- Chinese version will be used to measure stigma-related mental illness attitude of participants. MICA is a six-point scale that includes 16 items, and response options are from 1=totally agree to 6=totally disagree. The total score range is taken from 16-96. The internal consistency 66 is 0.72-0.75, and test-retest reliability is 0.76-0.87 of MICA in the Chinese version.A lower score indicates participants having a positive attitude towards schizophrenia.
Stigma behavior toward Schizophrenia as assessed by Reported and Intended Behavior Scale (RIBS) | up to three month
  Reported and Intended Behavior Scale (RIBS)-Chinese version will be used to measure the stigma-related mental illness behavior of participants. RIBS is a five-point scale that includes eight items, and response options are designed as 1=totally disagree, 2=disagree, 3=do not know, 4=agree, 5=totally agree. The total score range is taken from 4-20 of items 5-8. The internal consistency is 0.82, and test-retest reliability is 0.68 of RIBS in the Chinese version.The higher score indicates the participants are more willing to contact people who have schizophrenia.
Empathy toward Schizophrenia as assessed by Jefferson Scale of Empathy-Health Profession Students (JSE-HPS) | up to three month
  Jefferson Scale of Empathy-Health Profession Students (JSE-HPS)- Chinese version will be used to measure the nursing students' empathy towards people with schizophrenia. S-JSE-HPS is a seven-point scale that includes twenty items, and response options are designed as 1=totally disagree to 7= totally agree. The total score range is taken from 20-140. The internal consistency is 0.93, and test-retest reliability is 0.92 of JSE-HPS in the Chinese version.The higher score indicates the participants have greater empathic attitudes toward schizophrenia.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiang Ya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No
After finish this study

REFERENCES:
- [Background] Amini H, Shoar S, Tabatabaee M, Arabzadeh S. The Effect of Clinical Exposure to Patients on Medical Students' Attitude Towards Mental Illness. Iran J Psychiatry Behav Sci. 2016 May 10;10(3):e1887. doi: 10.17795/ijpbs-1887. eCollection 2016 Sep. PMID 27822275
- [Background] Amsalem D, Gothelf D, Dorman A, Goren Y, Tene O, Shelef A, Horowitz I, Dunsky LL, Rogev E, Klein EH, Mekori-Domachevsky E, Fischel T, Levkovitz Y, Martin A, Gross R. Reducing Stigma Toward Psychiatry Among Medical Students: A Multicenter Controlled Trial. Prim Care Companion CNS Disord. 2020 Feb 27;22(2):19m02527. doi: 10.4088/PCC.19m02527. PMID 32135042
- [Background] Angermeyer MC, Dietrich S. Public beliefs about and attitudes towards people with mental illness: a review of population studies. Acta Psychiatr Scand. 2006 Mar;113(3):163-79. doi: 10.1111/j.1600-0447.2005.00699.x. PMID 16466402
- [Background] Batson, C. D. (2009). These things called empathy: Eight related but distinct phenomena. In J. Decety & W. Ickes (Eds.), The social neuroscience of empathy (pp. 3-15). MIT Press. https://doi.org/10.7551/mitpress/9780262012973.003.0002
- [Background] Batson, C. D., Chang, J., Orr, R., & Rowland, J. (2002). Empathy, Attitudes, and Action: Can Feeling for a Member of a Stigmatized Group Motivate One to Help the Group? Personality and Social Psychology Bulletin, 28(12), 1656-1666. https://doi.org/10.1177/014616702237647
- [Background] Batson, C. D., Early, S., & Salvarani, G. (1997). Perspective Taking: Imagining How Another Feels Versus Imaging How You Would Feel. Personality and Social Psychology Bulletin, 23(7), 751-758. https://doi.org/10.1177/0146167297237008
- [Background] Borrelli B, Sepinwall D, Ernst D, Bellg AJ, Czajkowski S, Breger R, DeFrancesco C, Levesque C, Sharp DL, Ogedegbe G, Resnick B, Orwig D. A new tool to assess treatment fidelity and evaluation of treatment fidelity across 10 years of health behavior research. J Consult Clin Psychol. 2005 Oct;73(5):852-60. doi: 10.1037/0022-006X.73.5.852. PMID 16287385
- [Background] Brouwers EPM. Social stigma is an underestimated contributing factor to unemployment in people with mental illness or mental health issues: position paper and future directions. BMC Psychol. 2020 Apr 21;8(1):36. doi: 10.1186/s40359-020-00399-0. PMID 32317023
- [Background] Chen S, Zhang W, Zhang J. Stigma and schizophrenia. Lancet. 2009 Apr 18;373(9672):1335; author reply 1336-7. doi: 10.1016/S0140-6736(09)60764-9. No abstract available. PMID 19376440
- [Background] Corrigan PW, Morris SB, Michaels PJ, Rafacz JD, Rusch N. Challenging the public stigma of mental illness: a meta-analysis of outcome studies. Psychiatr Serv. 2012 Oct;63(10):963-73. doi: 10.1176/appi.ps.201100529. PMID 23032675
- [Background] Corrigan PW, Rao D. On the self-stigma of mental illness: stages, disclosure, and strategies for change. Can J Psychiatry. 2012 Aug;57(8):464-9. doi: 10.1177/070674371205700804. PMID 22854028
- [Background] Corrigan PW, River LP, Lundin RK, Penn DL, Uphoff-Wasowski K, Campion J, Mathisen J, Gagnon C, Bergman M, Goldstein H, Kubiak MA. Three strategies for changing attributions about severe mental illness. Schizophr Bull. 2001;27(2):187-95. doi: 10.1093/oxfordjournals.schbul.a006865. PMID 11354586
- [Background] Creswell, J. W. (2013). Qualitative Inquiry and Research Design: Choosing among Five Approaches (3rd ed.). SAGE Publications, Inc.
- [Background] Crisp AH, Gelder MG, Rix S, Meltzer HI, Rowlands OJ. Stigmatisation of people with mental illnesses. Br J Psychiatry. 2000 Jul;177:4-7. doi: 10.1192/bjp.177.1.4. PMID 10945080
- [Background] Demiroren, M., Saka, M., Senol, Y., Senturk, V., Baysal, O., & Oztuna, D. (2016). The Impact of Reflective Practices on Medical Students' Attitudes towards Mental Illness. Anatolian Journal of Psychiatry, 17(6), 466. https://doi.org/10.5455/apd.214188
- [Background] Dincer B, Inangil D. The effect of affective learning on alexithymia, empathy, and attitude toward disabled persons in nursing students: A randomized controlled study. Perspect Psychiatr Care. 2022 Apr;58(2):813-821. doi: 10.1111/ppc.12854. Epub 2021 May 24. PMID 34028038
- [Background] Duman ZC, Gunusen NP, Inan FS, Ince SC, Sari A. Effects of two different psychiatric nursing courses on nursing students' attitudes towards mental illness, perceptions of psychiatric nursing, and career choices. J Prof Nurs. 2017 Nov-Dec;33(6):452-459. doi: 10.1016/j.profnurs.2017.06.005. Epub 2017 Jun 22. PMID 29157575
- [Background] Foster, J. (2017). Mental Health Campaigns and Social Representations Theory: A Consideration. Papers on Social Representations, 26 (2), 4.1-4.21. https://doi.org/10.17863/CAM.28049
- [Background] Haddad M, Waqas A, Qayyum W, Shams M, Malik S. The attitudes and beliefs of Pakistani medical practitioners about depression: a cross-sectional study in Lahore using the Revised Depression Attitude Questionnaire (R-DAQ). BMC Psychiatry. 2016 Oct 18;16(1):349. doi: 10.1186/s12888-016-1069-1. PMID 27756274
- [Background] Haddad M, Waqas A, Sukhera AB, Tarar AZ. The psychometric characteristics of the revised depression attitude questionnaire (R-DAQ) in Pakistani medical practitioners: a cross-sectional study of doctors in Lahore. BMC Res Notes. 2017 Jul 27;10(1):333. doi: 10.1186/s13104-017-2652-3. PMID 28750688
- [Background] Hsiao CY, Tsai YF, Kao YC. Psychometric properties of a Chinese version of the Jefferson Scale of Empathy-Health Profession Students. J Psychiatr Ment Health Nurs. 2013 Dec;20(10):866-73. doi: 10.1111/jpm.12024. Epub 2012 Dec 4. PMID 23205565
- [Background] Hu, Y. Y. (2018, June). To Reduce Stigma in Patients with Schizophrenia in the Group Social Work Service South. Central University for Nationalities.
- [Background] Jorm AF, Reavley NJ, Ross AM. Belief in the dangerousness of people with mental disorders: a review. Aust N Z J Psychiatry. 2012 Nov;46(11):1029-45. doi: 10.1177/0004867412442406. Epub 2012 Mar 15. PMID 22422995
- [Background] Julious, S. A. (2005). Sample size of 12 per group rule of thumb for a pilot study. Pharmaceutical Statistics, 4(4), 287-291. https://doi.org/10.1002/pst.185
- [Background] Kassam A, Glozier N, Leese M, Loughran J, Thornicroft G. A controlled trial of mental illness related stigma training for medical students. BMC Med Educ. 2011 Jul 29;11:51. doi: 10.1186/1472-6920-11-51. PMID 21801355
- [Background] Li J, Li J, Thornicroft G, Huang Y. Levels of stigma among community mental health staff in Guangzhou, China. BMC Psychiatry. 2014 Aug 13;14:231. doi: 10.1186/s12888-014-0231-x. PMID 25115221
- [Background] Lincoln, Y. S., & Guba, E. G. (1986). But is it rigorous? Trustworthiness and authenticity in naturalistic evaluation. New Directions for Program Evaluation, 1986(30), 73-84. doi:10.1002/ev.1427
- [Background] Martin A, Chilton J, Gothelf D, Amsalem D. Physician Self-disclosure of Lived Experience Improves Mental Health Attitudes Among Medical Students: A Randomized Study. J Med Educ Curric Dev. 2020 Jan 8;7:2382120519889352. doi: 10.1177/2382120519889352. eCollection 2020 Jan-Dec. PMID 32363235
- [Background] Pan, S, M., Zhou Y., Luo, X, J., Feng, W, S., Lu, C, J., Lin, W, Q., Yan, X, S., Zhang, H., R, Y, X. (2013). Reliability and Validity of Chinese Version of Mental Illness：Clinician's Attitudes Scale. Chinese Journal of Practical Nursing, 29(33), 4-8.
- [Background] Papish A, Kassam A, Modgill G, Vaz G, Zanussi L, Patten S. Reducing the stigma of mental illness in undergraduate medical education: a randomized controlled trial. BMC Med Educ. 2013 Oct 24;13:141. doi: 10.1186/1472-6920-13-141. PMID 24156397
- [Background] Patten SB, Remillard A, Phillips L, Modgill G, Szeto ACh, Kassam A, Gardner DM. Effectiveness of contact-based education for reducing mental illness-related stigma in pharmacy students. BMC Med Educ. 2012 Dec 5;12:120. doi: 10.1186/1472-6920-12-120. PMID 23216787
- [Background] Reavley NJ, Jorm AF. The Australian public׳s beliefs about the causes of schizophrenia: associated factors and change over 16 years. Psychiatry Res. 2014 Dec 15;220(1-2):609-14. doi: 10.1016/j.psychres.2014.07.016. Epub 2014 Jul 16. PMID 25110311
- [Background] Sim J, Lewis M. The size of a pilot study for a clinical trial should be calculated in relation to considerations of precision and efficiency. J Clin Epidemiol. 2012 Mar;65(3):301-8. doi: 10.1016/j.jclinepi.2011.07.011. Epub 2011 Dec 9. PMID 22169081
- [Background] Suresh K. An overview of randomization techniques: An unbiased assessment of outcome in clinical research. J Hum Reprod Sci. 2011 Jan;4(1):8-11. doi: 10.4103/0974-1208.82352. PMID 21772732
- [Background] Taşkın, E. O., Özmen, D., Özmen, E., & Demet, M. M. (2003). Attitudes of School of Health Students towards Schizophrenia. Archives of Neuropsychiatry, 40(1), 5-12.
- [Background] Thornicroft G, Mehta N, Clement S, Evans-Lacko S, Doherty M, Rose D, Koschorke M, Shidhaye R, O'Reilly C, Henderson C. Evidence for effective interventions to reduce mental-health-related stigma and discrimination. Lancet. 2016 Mar 12;387(10023):1123-1132. doi: 10.1016/S0140-6736(15)00298-6. Epub 2015 Sep 22. PMID 26410341
- [Background] Tseng, W. (2013). Chinese Culture and Mental Health. Academic Press
- [Background] Tsimane TA, Downing C. Transformative learning in nursing education: A concept analysis. Int J Nurs Sci. 2019 Dec 16;7(1):91-98. doi: 10.1016/j.ijnss.2019.12.006. eCollection 2020 Jan 10. PMID 32099865
- [Background] Tsoi OYY, Chan SKW, Chui AHC, Hui CLM, Chang WC, Lee EHM, Henderson C, Chen EYH. Effect of brief social contact video compared with expert information video in changing knowledge and attitude towards psychosis patients among medical students. Early Interv Psychiatry. 2021 Apr;15(2):278-285. doi: 10.1111/eip.12938. Epub 2020 Feb 11. PMID 32043807
- [Background] Valery KM, Prouteau A. Schizophrenia stigma in mental health professionals and associated factors: A systematic review. Psychiatry Res. 2020 Aug;290:113068. doi: 10.1016/j.psychres.2020.113068. Epub 2020 May 24. PMID 32474069
- [Background] Van Daele T, Hermans D, Van Audenhove C, Van den Bergh O. Stress reduction through psychoeducation: a meta- analytic review. Health Educ Behav. 2012 Aug;39(4):474-85. doi: 10.1177/1090198111419202. Epub 2011 Oct 10. PMID 21986242
- [Background] Waqas A, Naveed S, Makhmoor A, Malik A, Hassan H, Aedma KK. Empathy, Experience and Cultural Beliefs Determine the Attitudes Towards Depression Among Pakistani Medical Students. Community Ment Health J. 2020 Jan;56(1):65-74. doi: 10.1007/s10597-019-00459-9. Epub 2019 Sep 11. PMID 31512078
- [Background] Waqas A, Zubair M, Ghulam H, Wajih Ullah M, Zubair Tariq M. Public stigma associated with mental illnesses in Pakistani university students: a cross sectional survey. PeerJ. 2014 Dec 16;2:e698. doi: 10.7717/peerj.698. eCollection 2014. PMID 25548734
- [Background] Wechsler D, Schomerus G, Mahlke C, Bock T. Effects of contact-based, short-term anti-stigma training for medical students : Results from a randomized controlled trial. Neuropsychiatr. 2020 Jun;34(2):66-73. doi: 10.1007/s40211-020-00337-x. Epub 2020 Feb 28. PMID 32112263
- [Background] Wittchen HU, Jacobi F, Rehm J, Gustavsson A, Svensson M, Jonsson B, Olesen J, Allgulander C, Alonso J, Faravelli C, Fratiglioni L, Jennum P, Lieb R, Maercker A, van Os J, Preisig M, Salvador-Carulla L, Simon R, Steinhausen HC. The size and burden of mental disorders and other disorders of the brain in Europe 2010. Eur Neuropsychopharmacol. 2011 Sep;21(9):655-79. doi: 10.1016/j.euroneuro.2011.07.018. PMID 21896369
- [Background] Yang LH. Application of mental illness stigma theory to Chinese societies: synthesis and new directions. Singapore Med J. 2007 Nov;48(11):977-85. PMID 17975685
- [Background] Yang LH, Chen FP, Sia KJ, Lam J, Lam K, Ngo H, Lee S, Kleinman A, Good B. "What matters most:" a cultural mechanism moderating structural vulnerability and moral experience of mental illness stigma. Soc Sci Med. 2014 Feb;103:84-93. doi: 10.1016/j.socscimed.2013.09.009. PMID 24507914
- [Background] Yang LH, Kleinman A. 'Face' and the embodiment of stigma in China: the cases of schizophrenia and AIDS. Soc Sci Med. 2008 Aug;67(3):398-408. doi: 10.1016/j.socscimed.2008.03.011. Epub 2008 Apr 15. PMID 18420325
- [Background] Yao, J., Cheng, Z., Su, Y, S. (2013). Advances in the Treatment of Refractory Schizophrenia. China Medical Herald. (10), 32-34.
- [Background] Zhou C, Li Z, Arthur D. Psychometric evaluation of the illness perception questionnaire for schizophrenia in a Chinese population. Asian J Psychiatr. 2020 Apr;50:101972. doi: 10.1016/j.ajp.2020.101972. Epub 2020 Feb 11. PMID 32109801
- [Derived] Chen X, Wang S, Liao X, Tam HL, Li Y, Leung SF, Bressington DT. A Chinese culture-specific intervention to decrease nursing students' stigma towards schizophrenia: a pilot feasibility randomised controlled trial. BMC Nurs. 2025 Aug 29;24(1):1130. doi: 10.1186/s12912-025-03743-0. PMID 40883707

DOCUMENTS (1):
  • Study Protocol (2022-02-24): https://cdn.clinicaltrials.gov/large-docs/08/NCT05413408/Prot_000.pdf